CLINICAL TRIAL: NCT06212856
Title: Effects of 8 Week Plyometric Training on Physical Fitness and Technical Skills in Young Male Volleyball Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 014245
Record Dates: First submitted 2023-12-26; First posted 2024-01-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Physical Fitness; Technical Skills
Keywords: Plyometric training; Young Male Volleyball Players; Physical fitness and technical skills
MeSH Terms: interventions — Plyometric Exercise; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Plyometric training) (Experimental)
  Interventions: Other: Plyometric training
- Group-B (Conventional) (Other)
  Interventions: Other: Conventional

INTERVENTIONS:
Other: Plyometric training — The group will receive plyometric exercises in a controlled environment. Following, Plyometrics would be performed.
  1. Leg hops
  2. Tuck jumps
  3. Vertical jumps
  4. Explosive push-ups
  5. Jumping spider
  6. Lateral/ diagonal and broad jumps
  7. Clapping push-ups
  8. Medicine ball presses
  9. Rotational throws
  10. Vertical and obstacle jumps
  11. Box shuffles
  12. Chest passes
  13. Box jumps
  14. Drop jumps
  15. Overarm throws
  Arms: Group-A (Plyometric training)
Other: Conventional — The group will receive conventional exercises in a controlled environment. Following, conventional exercises would be performed.
  1. Pushups.
  2. Situps.
  3. Lunges
  4. Squats
  5. 500m running
  Arms: Group-B (Conventional)

SUMMARY:
This study aims to find the effectiveness of Plyometric training on Physical fitness and Technical skills of young male volleyball players. Players would be taken from Prime Sports Academy and Prime Institute of Health Sciences, Islamabad and a well-designed Plyometric training plan will be implied on them for 8 weeks. After the time span, the result would be compared to check the effectiveness of the training plan.

DETAILED DESCRIPTION:
Volleyball, invented by William Morgan in 1895, boasts a global participation of approximately 500 million people, making it a dynamic and fast-paced sport with diverse technical, tactical, and athletic demands. The game places high requirements on players' speed, agility, power, and strength. In the Netherlands, it is one of the most played team sports, with over 12,500 athletes participating. Volleyball is considered safer than other sports like football, handball, and basketball. Plyometric training (PT) is a key focus for coaches and professionals aiming to enhance players' conditioning capacities.

Plyometric jump training (PJT) has been identified as beneficial for both amateur and professional volleyball players, emphasizing the importance of training for repeated jumping, frequent sprinting, and directional changes. A meta-analysis by Ramirez et al. (2020) found that PJT effectively improved players in various age groups and genders while being deemed safe for volleyball players. Gjinovci et al. (2017) conducted a Randomized Control Trial, revealing greater improvements in plyometric group participants compared to skill-based training, particularly for sprinting, jumping, and throwing performance in players above 18 years of age.

Given the lack of a structured training plan for volleyball players, the study proposes implementing a structured plyometric training plan. This approach aims to enhance physical fitness and technical skills, including improved landing mechanics, increased explosive power, muscle strength, and agility. The study anticipates incorporating the structured plyometric training plan into the domestic players' training protocol, with a focus on improving rate of force development (RFD) for explosive movements such as jumping and spiking, as well as enhancing speed and agility for quick and coordinated on-court actions. The ultimate goal is to evaluate whether the proposed training plan positively impacts players' technical skills and physical fitness.

ELIGIBILITY:
Inclusion Criteria:

* Young male healthy volleyball players aged 18-25 years, actively engaged in games for at least 6 months will be included in the study.

Exclusion Criteria:

* Female players
* History of trauma/injury in the last month.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 28 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-11-25 (Estimated)

PRIMARY OUTCOMES:
Vertical jumping test | 8 weeks
  Leg Power
Hand Dynamometer | 8 weeks
  Hand Strength
1RM test | 8 weeks
  Strength
30- Meter Sprint test. | 8 weeks
  Speed
W-agility test | 8 weeks
  Agility
2.4 km run test | 8 weeks
  Endurance Test
Sit and Reach test. | 8 weeks
  Flexibility
Abdominal Strength test. | 8 weeks
  Abdominal strength
Ruler drop test. | 8 weeks
  Reaction time
Medicine Ball Put Test | 8 weeks
Serving Test | 8 weeks
  * AAHPER Serving Test
  * AAHPERD Serving Test
BRUMBACH Serving Test | 8 weeks
Fore-arm Pass Test | 8 weeks
  * AAHPER Wall Volley
  * AAHPERD Pass-to-Self
Spiking Test | 8 weeks
  AAHPERD Wall Spike

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Prime Sports Academy & Prime Institute of Health Sciences, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No